CLINICAL TRIAL: NCT04778397
Title: A Phase 3, Randomized, Open-Label Study Evaluating the Safety and Efficacy of Magrolimab in Combination With Azacitidine Versus Physician's Choice of Venetoclax in Combination With Azacitidine or Intensive Chemotherapy in Previously Untreated Patients With TP53 Mutant Acute Myeloid Leukemia
Brief Title: Study of Magrolimab in Combination With Azacitidine Versus Physician's Choice of Venetoclax in Combination With Azacitidine or Intensive Chemotherapy in Patients With TP53 Mutant Acute Myeloid Leukemia That Have Not Been Treated
Acronym: ENHANCE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to futility.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-546-5857; 2020-003949-11 (EudraCT Number); jRCT2071220076 (Other: Japan Registry of Clinical Trials)
Expanded Access: NCT05627466 (No longer available)
Record Dates: First submitted 2021-02-23; First posted 2021-03-03 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — magrolimab; venetoclax; Azacitidine; Cytarabine; Daunorubicin; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Magrolimab + Azacitidine (Experimental): Participants will receive an escalating dose of magrolimab and a fixed dose of azacitidine.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- Control Arm: Venetoclax + Azacitidine (Active Comparator): Participants who are appropriate for non-intensive therapy will receive an escalating dose of venetoclax and a fixed dose of azacitidine.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Control Arm: 7+3 Chemotherapy (Active Comparator): Participants who are appropriate for intensive therapy will receive 7+3 chemotherapy: 7 day treatment with cytarabine and 3 day treatment with daunorubicin or idarubicin during induction and high-dose cytarabine and steroidal eye drops during consolidation.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Idarubicin; Drug: Steroidal Eye Drops

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously (IV).
  Other Names: GS-4721
  Arms: Magrolimab + Azacitidine
Drug: Venetoclax — Administered orally at a dose of 100 milligrams (mg) on Day 1, 200 mg on Day 2, 400 mg on Days 3-28 during Cycle 1, followed by 400 mg on Days 1-28 during every cycle (Cycle=28 days).
  Arms: Control Arm: Venetoclax + Azacitidine
Drug: Azacitidine — Administered either subcutaneously (SC) or IV, 75 milligrams per square meter (mg/m^2) on Days 1-7 or Days 1-5, 8 and 9 during every cycle (Cycle=28 days).
  Arms: Control Arm: Venetoclax + Azacitidine; Magrolimab + Azacitidine
Drug: Cytarabine — Induction: administered continuous infusion, 100 or 200 mg/m^2 on Days 1-7 (7+3 induction) and if needed Days 1-5 (5+2 induction) during a cycle (Cycle=Up to 42 Days).
  Consolidation: administered IV, 1500 or 3000 mg/m^2 on Days 1, 3, and 5 once every 12 hours for up to 4 cycles.
  Arms: Control Arm: 7+3 Chemotherapy
Drug: Daunorubicin — Administered IV peripherally (IVP), 60 mg/m^2 on Days 1-3 (7+3 induction) and if needed Days 1-2 (5+2 induction) during a cycle (Cycle=Up to 42 days).
  Arms: Control Arm: 7+3 Chemotherapy
Drug: Idarubicin — Administered IV, 12 mg/m^2 on Days 1-3 (7+3 induction) and if needed Days 1-2 (5+2 induction) during a cycle (Cycle=Up to 42 days).
  Arms: Control Arm: 7+3 Chemotherapy
Drug: Steroidal Eye Drops — Administered per institutional standard during consolidation.
  Arms: Control Arm: 7+3 Chemotherapy

SUMMARY:
The goal of this clinical study is to compare the effectiveness of the study drugs, magrolimab in combination with azacitidine, versus venetoclax in combination with azacitidine in participants with previously untreated TP53 mutant acute myeloid leukemia (AML).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with confirmation of acute myeloid leukemia (AML) by World Health Organization criteria, previously untreated for AML, and who have presence of at least 1 TP53 gene mutation that is not benign or likely benign based on evaluation by either central laboratory or an approved local laboratory (after central review of the bone marrow TP53 mitigation next-generation sequencing test results) (individuals with biallelic 17p deletions, loss of both 17p alleles, are eligible based on locally evaluated cytogenetics/karyotype/fluorescence in situ hybridization (FISH) report).
* Individuals with white blood cell (WBC) count ≤ 20×10^3/microliter (μL) prior to randomization. If the individual's WBC is > 20×10^3/μL prior to randomization, the individual can be enrolled, assuming all other eligibility criteria are met. However, the WBC should be ≤ 20×10^3/μL prior to the first dose of study treatment and prior to each magrolimab dose the first 4 weeks (if the individual is randomized to the experimental arm) Note: Individuals can be treated with hydroxyurea and/or leukapheresis throughout the study or prior to randomization to reduce the WBC to ≤ 20×10^3/μL to enable eligibility for study drug dosing.
* The hemoglobin must be ≥ 9 grams per deciliter (g/dL) prior to initial dose of study treatment.

Notes: Transfusions are allowed to meet hemoglobin eligibility.

* Individual has provided informed consent.
* Individual is willing and able to comply with clinic visits and procedure outlined in the study protocol.
* Individuals must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, except for individuals less than 75 years of age and appropriate for non-intensive treatment. For these individuals, the ECOG performance status score may be 0 to 3.
* Individuals must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 milliliters per minute calculated by the Cockcroft Gault formula.
* Adequate cardiac function as demonstrated by:

  * Lack of symptomatic congestive heart failure and clinically significant cardiac arrhythmias and ischemic heart disease.
  * Left ventricular ejection fraction (LVEF) > 50% for individuals appropriate for intensive therapy.
* Adequate liver function as demonstrated by:

  * Aspartate aminotransferase ≤ 3.0 × upper limit of normal (ULN).
  * Alanine aminotransferase ≤ 3.0 × ULN.
  * Total bilirubin ≤ 1.5 × ULN, or primary unconjugated bilirubin ≤ 3.0 × ULN if individual has a documented history of Gilbert's syndrome or genetic equivalent.
* Pretreatment blood cross-match completed.
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Individuals must be willing to consent to mandatory pretreatment and on-treatment bone marrow biopsies (aspirate and trephines).

Key Exclusion Criteria:

* Positive serum pregnancy test.
* Breastfeeding female.
* Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient.
* Prior treatment with any of the following:

  * Cluster of differentiation 47 (CD47) or signal regulatory protein alpha (SIRPα)-targeting agents
  * Antileukemic therapy for the treatment of AML (excluding hydroxyurea), hypomethylating agent (HMA), low dose cytarabine and/or venetoclax.

Note: Individuals with prior myelodysplastic syndrome (MDS) who have not received prior HMAs or chemotherapeutic agents for MDS are allowed on study. Other prior MDS therapies including, but not limited to, lenalidomide, erythroid stimulating agents, or similar red blood cell (RBC)-direct therapies, were allowed. Localized non-central nervous system (CNS) radiotherapy, erythroid and/or myeloid growth factors, hormonal therapy with luteinizing hormone-releasing hormone agonists for prostate cancer, hormonal therapy or maintenance for breast cancer, and treatment with bisphosphonates and receptor activator of nuclear factor kappa-B ligand inhibitors are also not criteria for exclusion.

* Individuals who are appropriate for intensive treatment but who have been previously treated with maximum cumulative doses of idarubicin and/or other anthracyclines and anthracenediones will be excluded.
* Individuals receiving any live vaccine within 4 weeks prior to initiation of study treatments.
* For individuals appropriate for intensive therapy, individuals treated with trastuzumab within 7 months prior to initiation of study treatments.
* Current participation in another interventional clinical study.
* Known inherited or acquired bleeding disorders.
* Individuals appropriate for non-intensive therapy, who have received treatment with strong and/or moderate cytochrome P450 enzyme 3A (CYP3A) inducers within 7 days prior to the initiation of study treatments.
* Individuals appropriate for non-intensive therapy who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or starfruit within 3 days prior to the initiation of study treatment.
* Individuals appropriate for non-intensive therapy who have malabsorption syndrome or other conditions that preclude enteral route of administration.
* Clinical suspicion of active CNS involvement with AML.
* Individuals who have acute promyelocytic leukemia.
* Significant disease or medical conditions, as assessed by the investigator and sponsor, that would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV.
* Second malignancy, except MDS, treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which individuals are not on active anti-cancer therapies and have had no evidence of active malignancy for at least ≥ 1 year Note: Individuals on maintenance therapy alone who have no evidence of active malignancy for at least ≥ 1 year are eligible.
* Known active or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or human immunodeficiency virus (HIV) infection in medical history.
* Active HBV, and/or active HCV, and/or HIV following testing at screening:

  * Individuals who test positive for hepatitis B surface antigen (HBsAg). Individuals who test positive for hepatitis B core antibody (anti-HBc) will require HBV deoxyribose nucleic acid (DNA) by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
  * Individuals who test positive for HCV antibody. These individuals will require HCV ribose nucleic acid (RNA) quantitative PCR for confirmation of active disease.
  * Individuals who test positive for HIV antibody.
  * Individuals not currently receiving antiviral therapy and who have an undetectable viral load in the prior 3 months may be eligible for the study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (156):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - USC/ Norris Comprehensive Cancer Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Irvine Health, Orange, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital/Main Lab, Chicago, Illinois
  - The University of Chicago Medical Centre, Chicago, Illinois
  - University of Kansas Hospital, Fairway, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Tulane Medical center, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center Outpatient Pharmacy, Rochester, Minnesota
  - MidAmerica Division, Inc., c/o Research Medical Center, Kansas City, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Blood Cancer Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center/ James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Research Organization, Philadelphia, Pennsylvania
  - St. Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Baylor College of Medicine Medical Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute ,The University of Utah, Salt Lake City, Utah
  - Froedtert Hospital / Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (10):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Calvary Master Newcastle, Waratah, New South Wales
  - Westmead Hospital / Department of Haematology and Bone Marrow Transplantation, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Andrew Love Cancer Centre, University Hospital Geelong, Geelong, Victoria
  - The Alfred, Melbourne, Victoria
  - St Vincents Hospital Melbourne, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Univ. -Klinik für Hämatologie und Internistische Onkologie, Kepler Universitätskilkun GmbHMed, Linz
  - Uniklinikum Salzburg, Universitatsklinik f. Innere Medizin III der PMU, Salzburg
- Belgium (6):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende AV, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Grand Hôpital De Charleroi - Notre Dame, Charleroi
  - Universitaire Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Delta vzw, Roeselare
- Canada (6):
  - Tom Baker Cancer Center, Calgary
  - Queen Elizabeth II Health Sciences Centre, Halifax
  - CIUSSS de L'Est-de-L'Ile-de- Montreal - Hopital Maisonneuve-Rosemont, Montreal
  - McGill University Health Centre, Montreal
  - Sunnybrook Research Institute, Toronto
  - Princess Margaret Cancer Centre, Toronto
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense C
- France (12):
  - CHU d'Angers, Angers
  - CHU de Caen, Caen
  - CHRU Lille - Hospital Claude Huriez, Lille
  - CHU Limoges, Limoges
  - Central Hospital Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes, Hotel Dieu, Nantes
  - CHU Nice - Hopital Archet 1, Nice
  - Gustave Roussy, Paris
  - Hopital Haut-Leveque, Pessac
  - IUCT Oncopole, Toulouse
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (13):
  - Uniklinik RWTH Aachen, Medizinische Klunuk IV - Klinik fur Hamatologie, Onkologie, Hamastaseologie und Srammzelltransplantation, Aachen
  - Dept. of Hematology, Oncology and Tumor Immunology, Charite- University Medicine Berlin, Campus Virchow Klinikum, Berlin
  - Department of Hematology and Oncology, Braunschweig Community Hospital, Braunschweig
  - Universitatsklinikum Koln, Cologne
  - Universitatsklinikum Carl Gustav Carus Dresden an der Technische Universitat Dresden, Medizinische Klinik und Poliklinik 1, Bereich Hamatologie, Dresden
  - Universitätsklinikum Düsseldorf -Klinik für Hämatologie, Onkologie und Klinische Immunologie, Düsseldorf
  - Dept. of Medicine II, University Hospital Hamburg-Eppendorf, Hamburg
  - Universitatsklinikum Heidelberg, Innere Medizin V, Hamatologie, Onkologie und Rheumatologie, Heidelberg
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Klinikum Ludwigshafen Medizinische Klinik A, Ludwigshafen
  - LMU - Klinikum der Universitat Munchen, Medizinische Klinik und Poliklinik III, Campus Grosshadern, München
  - Klinikum rechts der Isar der Technischen Universitat Munchen, Klinik und Poliklinik fur Innere Medizin III, München
  - Universitatsklinikum Ulm, Zentrum fur Innere Medizin, Innere Medizin III, Ulm
- Hong Kong (2):
  - Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Italy (10):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - AOU Consorziale Policlinico Bari, Bari
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant'Orsola-Malphigi U.O Ematologia, Bologna
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRS - Oncologia Medica, Meldola
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli U.O.S.C. di Ematologia con Trapianto di Midollo Osseo, Napoli
  - SC Ematologia, Azienda Ospedaliera di Perugia - Santa Maria della Misericordia, Perugia
  - AORM - AO Riuniti Marche Norde - Pesaro Presidio "San Salvatore" - Muraglia, Pesaro
  - Fondazione PTV Policinico Tor Vergata, Roma
  - SCDU Ematologia e Terrapie cellulari AO O Ordine Mauriziano Torino, Torino
  - ASST Sette Laghi - Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (23):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki
  - Chiba Aoba Municipal Hospital, Chiba
  - University of Yamanashi Hospital, Chūō
  - Kyushu University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Aiiku Hospital, Hokkaido
  - Tokai University School of Medicine, Isehara
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi
  - Ehime Prefectural Center Hospital, Matsuyama
  - Nagasaki University Hospital, Nagasaki
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Kindai University Hospital, Sayama
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai
  - NTT Medical Center Tokyo, Shinagawa-Ku
  - Yamagata University Hospital, Yamagata
  - University of Fukui Hospital, Yoshida-gun
- Spain (19):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Complejo Asistencial Universitario de Burgos/H.U. de Burgos, Burgos
  - Complejo Hospitalario San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Clinica Universidad de Navarra - Pamplona (Main Site), Pamplona
  - Complejo Asistencial Universitario de Salamanca - Hsopital Clinico, Salamanca
  - Hospital U. Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari I Politècnic La Fe, Valencia
- Universitetssjukhus, Hematologimottagnungen, Lund, Sweden
- Switzerland (2):
  - Universitatsspital Basel - Klinik fur Hamatrologie, Bereich Innere Medizin, Basel
  - Inselspital, Universitatsspital Bern - Universitatsklinik fur Medizinisch Onkologie, Bern
- United Kingdom (12):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - United Lincolnshire Hospitals NHS Trust, Pilgrim Hospital, Sibsey Road, Boston
  - Cambridge University Hospital NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff Wales
  - Barts Health NHS Trust, City of London
  - NHS Tayside, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - King's College NHS Foundation Trust, London
  - Oxford University Hospital NHS Foundation Trust, Oxford
  - The Royal Marsden NHS Foundation Trust, Sutton
  - The Christie NHS Foundation Trust, Withington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeidner JF, Sallman DA, Recher C, Daver NG, Leung AYH, Hiwase DK, Subklewe M, Pabst T, Montesinos P, Larson RA, Wilde L, Enjeti AK, Kawashima I, Papayannidis C, O'Nions J, Johnson L, Dong M, Huang J, Bagheri T, Hacohen Kleiman G, Lee C, Vyas P. Magrolimab plus azacitidine vs physician's choice for untreated TP53-mutated acute myeloid leukemia: the ENHANCE-2 study. Blood. 2025 Jul 31;146(5):590-600. doi: 10.1182/blood.2024027408. PMID 40009500
- [Derived] Daver NG, Vyas P, Kambhampati S, Al Malki MM, Larson RA, Asch AS, Mannis G, Chai-Ho W, Tanaka TN, Bradley TJ, Jeyakumar D, Wang ES, Sweet K, Kantarjian HM, Garcia-Manero G, Komrokji R, Xing G, Ramsingh G, Renard C, Zeidner JF, Sallman DA. Tolerability and Efficacy of the Anticluster of Differentiation 47 Antibody Magrolimab Combined With Azacitidine in Patients With Previously Untreated AML: Phase Ib Results. J Clin Oncol. 2023 Nov 1;41(31):4893-4904. doi: 10.1200/JCO.22.02604. Epub 2023 Sep 13. PMID 37703506
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-546-5857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 841 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in North America, the United Kingdom, Europe, Asia, and, Australia. 1 participant was enrolled but was not randomized.
Groups:
- Magrolimab + Azacitidine (Non-Intensive Therapy): Participants who were appropriate for non-intensive therapy received 1 mg/kg magrolimab intravenously (IV) on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then every week (QW) x 5 weekly 30 mg/kg dose; 30 mg/kg every 2 weeks (Q2W) beginning 1 week after the 5 weekly 30 mg/kg dose. Participants received azacitidine subcutaneously (SC) or IV, 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9 during every cycle of 28 days. The treatment duration was up to a maximum of 1.3 years.
- Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy): Participants who were appropriate for non-intensive therapy received Venetoclax 100 mg orally on Cycle 1 Day 1; 200 mg orally on Cycle 1 Day 2; 400 mg orally on Cycle 1 Day 3 everyday and throughout all the cycles. Participants received azacitidine SC or IV, 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9 during every cycle of 28 days. The treatment duration was up to a maximum of 1.3 years.
- Magrolimab + Azacitidine (Intensive Therapy): Participants who were appropriate for intensive therapy received 1 mg/kg magrolimab IV on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 weekly 30 mg/kg dose; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose. Participants received azacitidine SC or IV, 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9 during every cycle of 28 days. The treatment duration was up to a maximum of 1.3 years.
- Control Arm: 7+3 Chemotherapy (Intensive Therapy): Participants who were appropriate for intensive therapy received 7+3 chemotherapy: 7 day treatment with cytarabine 100 or 200 mg/m^2 continuous infusion and 3 day treatment with daunorubicin 60 mg/m^2 IV push or idarubicin 60 mg/m^2 IV during induction and high-dose cytarabine 1500 or 3000 mg/m^2 IV every 12 hours on Days 1, 3, and 5 up to 4 cycles and steroidal eye drops during consolidation. Each cycle was 28 days.
Period: Overall Study
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) | Magrolimab + Azacitidine (Intensive Therapy) | Control Arm: 7+3 Chemotherapy (Intensive Therapy)
Started | 101 | 104 | 27 | 25
Completed | 0 | 0 | 0 | 0
Not Completed | 101 | 104 | 27 | 25
Not completed — Death | 59 | 54 | 11 | 9
Not completed — Study Terminated by Sponsor | 34 | 42 | 15 | 12
Not completed — Withdrew Consent | 5 | 4 | 1 | 1
Not completed — Reason Not Specified | 1 | 3 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat Analysis Set included all participants who were randomized in the study, with treatment assignment designated according to the treatment arm the participant was randomized to.
Groups:
- Magrolimab + Azacitidine (Non-Intensive Therapy): Participants who were appropriate for non-intensive therapy received 1 mg/kg magrolimab intravenously (IV) on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 weekly 30 mg/kg dose; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose. Participants received azacitidine subcutaneously (SC) or IV, 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9 during every cycle of 28 days. The treatment duration was up to a maximum of 1.3 years.
- Control Arm: 7+3 Chemotherapy (Intensive Therapy): Participants who were appropriate for intensive therapy received 7+3 chemotherapy: 7 day treatment with cytarabine 100 or 200 mg/m^2 continuous infusion and 3 day treatment with daunorubicin 60 mg/m^2 IV push or idarubicin 60 mg/m^2 IV during induction and high-dose cytarabine 1500 or 3000 mg/m^2 IV every 12 hours on Days 1, 3, and 5 up to 4 cycles and steroidal eye drops during consolidation up to 32 months. Each cycle was 28 days.
- Total: Total of all reporting groups
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) | Magrolimab + Azacitidine (Intensive Therapy) | Control Arm: 7+3 Chemotherapy (Intensive Therapy) | Total
Number analyzed (Participants) | 101 | 104 | 27 | 25 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 23 | 21 | 15 | 78
  >=65 years | 82 | 81 | 6 | 10 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9.6) | 71 (8.0) | 57 (9.6) | 61 (8.6) | 68 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 5 | 11 | 102
  Male | 58 | 61 | 22 | 14 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 1 | 2 | 25
  Not Hispanic or Latino | 82 | 74 | 19 | 20 | 195
  Unknown or Not Reported | 10 | 17 | 7 | 3 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 11 | 3 | 4 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 2 | 2 | 2 | 0 | 6
  White | 75 | 72 | 12 | 15 | 174
  More than one race | 4 | 2 | 1 | 2 | 9
  Unknown or Not Reported | 8 | 17 | 8 | 4 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 33 | 1 | 0 | 65
  Spain | 10 | 10 | 6 | 9 | 35
  France | 6 | 13 | 7 | 6 | 32
  United Kingdom | 12 | 11 | 2 | 1 | 26
  Australia | 5 | 7 | 4 | 4 | 20
  Japan | 8 | 9 | 2 | 2 | 21
  Italy | 7 | 10 | 1 | 0 | 18
  Germany | 9 | 5 | 0 | 2 | 16
  Switzerland | 5 | 2 | 1 | 0 | 8
  Hong Kong | 4 | 1 | 0 | 0 | 5
  Belgium | 1 | 1 | 2 | 0 | 4
  Canada | 2 | 0 | 1 | 1 | 4
  Austria | 1 | 1 | 0 | 0 | 2
  Sweden | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants Appropriate for Non-intensive Therapy
Description: OS was measured from the date of randomization to the date of death from any cause. Deaths which were not observed during the study were censored at their last known alive date.
  Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 2.1 years
Population: Participants from the Intent-to-Treat Analysis (ITT) Set who were appropriate for non-intensive therapy were analyzed. As per the pre-specified analysis, the data in this outcome measure was reported only for the non-intensive therapy groups.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy)
Number analyzed (Participants) | 101 | 104
months | 4.4 [3.6 to 6.0] | 6.6 [4.8 to 8.1]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine (Non-Intensive Therapy) vs Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy); Test type: Superiority; p = 0.5070, Stratified log-rank test; P-value from stratified log-rank test; Stratified Hazard Ratio = 1.132, 95% CI 2-sided [0.783 to 1.637]; Hazard ratio and 95% CIs were calculated using the Cox proportional hazards model, adjusted for randomization stratification factors (appropriateness for non-intensive therapy vs intensive therapy, age (< 75 years, >=75 years), geographic region (US sites, outside the US sites))

2. Secondary Outcome: Overall Survival in All Participants
Description: OS was measured from the date of randomization to the date of death from any cause. Deaths which were not observed during the study were censored at their last known alive date.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2.1 years
Population: Participants from the Intend-To-Treat Analysis Set were analyzed. As per the pre-specified analysis, the data for this outcome measure were analyzed together for all participants who received magrolimab + azacitidine and participants who received venetoclax + azacitidine or 7+3 chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Magrolimab + Azacitidine: Participants who were appropriate for intensive and non-intensive therapy received 1 mg/kg magrolimab intravenously (IV) on Days 1, 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, and then QW x 5 weekly 30 mg/kg dose; 30 mg/kg Q2W beginning 1 week after the 5 weekly 30 mg/kg dose. Participants received azacitidine subcutaneously (SC) or IV, 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9 during every cycle of 28 days. The treatment duration was up to a maximum of 1.3 years.
- Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy: Participants who were appropriate for non-intensive therapy received Venetoclax 100 mg orally on Cycle 1 Day 1; 200 mg orally on Cycle 1 Day 2; 400 mg orally on Cycle 1 Day 3 everyday and throughout all the cycles. Participants received azacitidine SC or IV, 75 mg/m^2 on Days 1-7 or Days 1-5, 8 and 9 during every cycle of 28 days. The treatment duration was up to a maximum of 1.3 years.
  Participants who were appropriate for intensive therapy received 7+3 chemotherapy: 7 day treatment with cytarabine 100 or 200 mg/m^2 continuous infusion and 3 day treatment with daunorubicin 60 mg/m^2 IV push or idarubicin 60 mg/m^2 IV during induction and high-dose cytarabine 1500 or 3000 mg/m^2 IV every 12 hours on Days 1, 3, and 5 up to 4 cycles and steroidal eye drops during consolidation. Each cycle was 28 days.
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 128 | 129
months | 4.4 [3.7 to 6.6] | 6.6 [4.9 to 8.9]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy; Test type: Superiority; p = 0.3237, Stratified Log-rank test; P-value from stratified log-rank test; Stratified Hazard Ratio = 1.183, 95% CI 2-sided [0.845 to 1.654]; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Event-Free Survival (EFS) in All Participants
Description: EFS: time from randomization to earliest relapse from CR (CR without minimal residual disease (CRMRD-) and CR with MRD positive/MRD unknown (CRMRD+/unk)), treatment failure (failure to achieve CR in 6 months of magrolimab/venetoclax+azacitidine; 2 months after chemotherapy), or death within the response window. CRMRD- and CRMRD+/unk: neutrophils >1.0 ×10^9/L, platelets >100 ×10^9/L, <5% bone marrow blasts, no circulating blasts or extramedullary disease (confirmed by flow cytometry <0.1% sensitivity for CRMRD-). Post-SCT assessments or new AML therapies were included. Date of randomization was assigned as event date for participants with treatment failure. Participants without events were censored at their last assessment. KM estimates were used for analysis.
Time Frame: Up to 2.1 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 128 | 129
months | 0.0 [NA to NA] — Upper and lower limits of the confidence interval (CI) could not be estimated due to a limitation in the Kaplan-Meier model, as the EFS values were below the level of quantification for this outcome measure. | 0.0 [NA to NA] — Upper and lower limits of the confidence interval (CI) could not be estimated due to a limitation in the Kaplan-Meier model, as the EFS values were below the level of quantification for this outcome measure.
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy; Test type: Superiority; p = 0.0661, Stratified Log-rank test; P-value for comparing the event free survival functions from the two treatment groups was from stratified log-rank test, adjusted for randomization; Stratified Hazard Ratio = 1.389, 95% CI 2-sided [1.043 to 1.848]; Hazard ratio and 95% CIs were calculated using the Cox proportional hazards model, adjusted for randomization stratification factors: therapy appropriateness, age (< 75 years, >=75 years), geographic region (US sites, outside the US sites)

4. Secondary Outcome: Rate of Complete Remission (CR) in All Participants
Description: The rate of CR was the percentage of participants who achieved a CR, including CR without minimal residual disease (CR MRD-) and CR with positive or unknown minimal residual disease (CR MRD+/unk) within 6 months of treatment with magrolimab + azacitidine or venetoclax + azacitidine, or within 2 months of treatment with 7 + 3 chemotherapy, as defined by investigators based on European Leukemia Net (ELN) 2017 AML (ELN 2017 AML) with modifications, while on study prior to initiation of any new anti-AML therapy or stem cell transplant (SCT) within the response assessment window of 2.1 years. CR MRD- and CR MRD+/unk are defined in Outcome Measure#3 (EFS). Percentages were rounded-off.
  Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 2.1 years
Population: Participants from the Intent-To-Treat Analysis Set were analyzed. As per the pre-specified analysis, the data for this outcome measure were analyzed together for all participants who received magrolimab + azacitidine and participants who received venetoclax + azacitidine or 7+3 chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 128 | 129
percentage of participants | 9.4 [4.9 to 15.8] | 29.5 [21.8 to 38.1]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy; Test type: Superiority; Stratified Odds Ratio = 0.250, 95% CI 2-sided [0.123 to 0.506]; Odds ratio and 2-sided 95% CI were calculated from stratum-adjusted Mantel-Haenszel estimates adjusted for randomization stratification factors (appropriateness for non-intensive therapy versus intensive therapy, age (< 75 years, >=75 years), geographic region (US sites, outside US sites))

5. Secondary Outcome: Rate of CR Without Minimal Residual Disease (CR MRD-) in All Participants
Description: Rate of CR MRD- was the percentage of participants who achieve a CR MRD- within 6 months treatment with magrolimab + azacitidine or venetoclax + azacitidine, or within 2 months of treatment with 7 + 3 chemotherapy, as defined by investigators based on ELN 2017 AML with modifications, while on study prior to initiation of any new anti-AML therapy or SCT within the response assessment window of 2.1 years. CR MRD- is defined in Outcome Measure #3 (EFS). Percentages were rounded-off.
  Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 2.1 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 128 | 129
percentage of participants | 0.8 [0.0 to 4.3] | 10.1 [5.5 to 16.6]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy; Test type: Superiority; Stratified Odds Ratio = 0.072, 95% CI 2-sided [0.009 to 0.559]; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Rate of CR and CR With Partial Hematologic Recovery (CR+CRh) in All Participants
Description: The CR+CRh rate was the percentage of participants who achieved a CR (including CR MRD- and CR MRD+/unk) or CRh as defined by CR with partial platelet and absolute neutrophil count (ANC) recovery within 6 months of treatment with magrolimab + azacitidine or venetoclax + azacitidine, or within 2 months of treatment with 7 + 3 chemotherapy while on study prior to initiation of any new anti-AML therapy or SCT up to the response assessment window of 2.1 years. CRh is defined as neutrophils > 0.5 x 10^9/L; platelets > 50 x 10^9/L; bone marrow blasts < 5%; Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease. CR MRD- and CR MRD+/unk are defined in Outcome Measure#3 (EFS). Percentages were rounded-off.
  Clopper-Pearson method were used in outcome measure analysis.
Time Frame: Up to 2.1 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 128 | 129
percentage of participants | 10.2 [5.5 to 16.7] | 34.1 [26.0 to 43.0]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy; Test type: Superiority; Stratified Odds Ratio = 0.215, 95% CI 2-sided [0.108 to 0.428]; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: Duration of CR (DCR)
Description: DCR was measured from the time the assessment criteria were first met for CR (including CR MRD- and CR MRD+/unk) within 6 months of treatment with magrolimab + azacitidine or venetoclax + azacitidine, or within 2 months of treatment with 7 + 3 chemotherapy, until the first date of AML relapse or death (including assessments post SCT). Participants who were not observed to have relapsed disease or death while on study were censored at the date of their last response assessment with no evidence of relapse. Participants who started taking new anti-AML therapies (excluding post-SCT maintenance therapy) before relapse, the DCR were censored at the last response assessment before the initiation of the new anti-AML therapies. CR MRD- and CR MRD+/unk are defined in Outcome Measure#3 (EFS).
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 2.1 years
Population: Participants from the Intent-To-Treat Analysis Set who achieved CR within 6 months in all participants (2 months for participants receiving 7 + 3 chemotherapy) were analyzed. As per the pre-specified analysis, the data for this outcome measure were analyzed together for all participants who received magrolimab + azacitidine and participants who received venetoclax + azacitidine or 7+3 chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 12 | 38
months | 9.5 [2.0 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 4.9 [3.1 to 6.5]

8. Secondary Outcome: Duration of CR+CRh
Description: Duration of CR+CRh was measured from the time the assessment criteria were first met for CR (including CR MRD- and CR MRD+/unk) or CRh within 6 months of treatment with magrolimab + azacitidine or venetoclax + azacitidine, or within 2 months of treatment with 7 + 3 chemotherapy, until the first date of AML relapse or death (including assessments post SCT). Participants who were not observed to have relapsed disease or death while on study were censored at the date of their last response assessment with no evidence of relapse. Participants who started taking new anti-AML therapies (excluding post-SCT maintenance therapy) before relapse, the duration of CR + CRh were censored at the last response assessment before the initiation of the new anti-AML therapies. CR MRD- and CR MRD+/un are defined in Outcome Measure #3. CRh is defined in Outcome Measure #6.
  KM estimates were used for outcome measure analysis.
Time Frame: Up to 2.1 years
Population: Participants from the Intent-To-Treat Analysis Set with who achieved CR+CRh within 6 months in all participants (2 months for participants receiving 7 + 3 chemotherapy) were analyzed. As per the pre-specified analysis, the data for this outcome measure were analyzed together for all participants who received magrolimab + azacitidine and participants who received venetoclax + azacitidine or 7+3 chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Control Arm: Venetoclax + Azacitidine or 7+3 Chemotherapy
Number analyzed (Participants) | 13 | 44
months | 9.5 [2.0 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events. | 4.9 [3.1 to 6.5]

9. Secondary Outcome: Percentage of Participants Experiencing Grade ≥ 3 Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any AE that began on or after the date of first dose of study treatment up to the date of last dose of study treatment plus 70 days or the day before initiation of new anti-AML therapy including SCT, whichever occurred first. Percentages were rounded-off.
Time Frame: First dose date up to 1.3 years plus 70 days
Population: The Safety Analysis Set included all participants who took at least 1 dose of any study treatment, with treatment assignment designated according to the actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) | Magrolimab + Azacitidine (Intensive Therapy) | Control Arm: 7+3 Chemotherapy (Intensive Therapy)
Number analyzed (Participants) | 96 | 98 | 27 | 23
percentage of participants | 96.9 | 95.9 | 92.6 | 95.7

10. Secondary Outcome: Percentage of Participants Experiencing Grade 3 or 4 Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study treatment plus 70 days or the day before initiation of any new anti-AML therapy including SCT, whichever occurred first. Percentages were rounded-off.
Time Frame: First dose date up to 1.3 years plus 70 days
Population: Participants from Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) | Magrolimab + Azacitidine (Intensive Therapy) | Control Arm: 7+3 Chemotherapy (Intensive Therapy)
Number analyzed (Participants) | 96 | 98 | 27 | 23
percentage of participants | 96.9 | 99.0 | 100 | 95.7

11. Secondary Outcome: Serum Concentration of Magrolimab
Time Frame: Predose on Days 1, 4, 8, 11; Days 29 and 57 Predose and 1 hour Postdose; Predose on Days 113, 169, 253, 281 and 337
Population: The Pharmacokinetic (PK) Analysis Set included all randomized participants who took at least one dose of magrolimab and have at least 1 measurable (non-below the limit of quantitation (BLQ) numeric values) posttreatment serum concentration of magrolimab. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Magrolimab + Azacitidine
Number analyzed (Participants) | 88
μg/mL
  Day 1 Predose | 0.0 (0.0)
  Day 4 Predose: number analyzed (Participants) | 1
  Day 4 Predose | 0.0 (NA) — Standard deviation cannot be calculated for 1 participant.
  Day 8 Predose: number analyzed (Participants) | 83
  Day 8 Predose | 0.0 (0.0)
  Day 11 Predose: number analyzed (Participants) | 1
  Day 11 Predose | 111 (NA) — Standard deviation cannot be calculated for 1 participant.
  Day 29 Predose: number analyzed (Participants) | 69
  Day 29 Predose | 311 (195)
  Day 29 1 hour Postdose: number analyzed (Participants) | 1
  Day 29 1 hour Postdose | 376 (NA) — Standard deviation cannot be calculated for 1 participant.
  Day 57 Predose: number analyzed (Participants) | 43
  Day 57 Predose | 402 (262)
  Day 57 1 hour Postdose: number analyzed (Participants) | 36
  Day 57 1 hour Postdose | 967 (351)
  Day 113 Predose: number analyzed (Participants) | 20
  Day 113 Predose | 138 (96.0)
  Day 169 Predose: number analyzed (Participants) | 10
  Day 169 Predose | 198 (129)
  Day 253 Predose: number analyzed (Participants) | 8
  Day 253 Predose | 294 (181)
  Day 281 Predose: number analyzed (Participants) | 1
  Day 281 Predose | 263 (NA) — Standard deviation cannot be calculated for 1 participant.
  Day 337 Predose: number analyzed (Participants) | 3
  Day 337 Predose | 251 (114)

12. Secondary Outcome: Percentage of Participants With Anti-Magrolimab Antibodies
Description: Percentages were rounded-off.
Time Frame: Up to 2 years
Population: The Immunogenicity Analysis Set included all randomized participants who received at least one dose of magrolimab and had at least one evaluable anti-magrolimab antibody test result.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Magrolimab + Azacitidine (Intensive Therapy)
Number analyzed (Participants) | 93 | 27
percentage of participants | 10.4 | 11.1

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 2.1 years; Adverse events: Up to 1.3 years plus 70 days
Description: All-cause mortality: The Intent-To-Treat Analysis Set included all participants who were randomized in the study, with treatment assignment designated according to the treatment arm the participant was randomized to.
  Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study treatment, with treatment assignment designated according to the actual treatment received.
Arm/Group | Magrolimab + Azacitidine (Non-Intensive Therapy) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) | Magrolimab + Azacitidine (Intensive Therapy) | Control Arm: 7+3 Chemotherapy (Intensive Therapy)
All-Cause Mortality (participants affected / at risk) | 61/101 | 57/104 | 14/27 | 10/25
Serious Adverse Events (participants affected / at risk) | 84/96 | 76/98 | 20/27 | 14/23
Other Adverse Events (participants affected / at risk) | 92/96 | 94/98 | 27/27 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab + Azacitidine (Non-Intensive Therapy) (N=96) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) (N=98) | Magrolimab + Azacitidine (Intensive Therapy) (N=27) | Control Arm: 7+3 Chemotherapy (Intensive Therapy) (N=23)
Anaemia (Blood and lymphatic system disorders) | 9 | 0 | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 32 | 34 | 7 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Red blood cell abnormality (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Orbital haematoma (Eye disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal vascular thrombosis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Device related thrombosis (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 1 | 1 | 1
Pyrexia (General disorders) | 10 | 4 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 1 | 0
Anal fistula infection (Infections and infestations) | 1 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 1 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Clostridial sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 3 | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 3 | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 13 | 10 | 2 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 2 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Rhinocerebral mucormycosis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 7 | 5 | 3 | 3
Septic shock (Infections and infestations) | 2 | 4 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 3 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab + Azacitidine (Non-Intensive Therapy) (N=96) | Control Arm: Venetoclax + Azacitidine (Non-Intensive Therapy) (N=98) | Magrolimab + Azacitidine (Intensive Therapy) (N=27) | Control Arm: 7+3 Chemotherapy (Intensive Therapy) (N=23)
Anaemia (Blood and lymphatic system disorders) | 25 | 28 | 7 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 25 | 7 | 11
Haemolysis (Blood and lymphatic system disorders) | 7 | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 26 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 16 | 3 | 5
Atrial fibrillation (Cardiac disorders) | 5 | 6 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 6 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 4 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 11 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6 | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 33 | 37 | 13 | 4
Diarrhoea (Gastrointestinal disorders) | 27 | 38 | 5 | 9
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 6 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 5 | 8 | 3 | 1
Nausea (Gastrointestinal disorders) | 27 | 32 | 11 | 6
Proctalgia (Gastrointestinal disorders) | 0 | 8 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 15 | 3 | 6
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 15 | 22 | 4 | 1
Asthenia (General disorders) | 13 | 13 | 3 | 1
Chills (General disorders) | 9 | 4 | 0 | 0
Fatigue (General disorders) | 24 | 20 | 2 | 0
Generalised oedema (General disorders) | 2 | 1 | 2 | 2
Injection site reaction (General disorders) | 5 | 15 | 3 | 0
Mucosal inflammation (General disorders) | 3 | 2 | 2 | 1
Non-cardiac chest pain (General disorders) | 3 | 5 | 0 | 0
Oedema (General disorders) | 3 | 0 | 1 | 6
Oedema peripheral (General disorders) | 17 | 19 | 4 | 6
Pyrexia (General disorders) | 40 | 24 | 11 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 6 | 2 | 0
Furuncle (Infections and infestations) | 0 | 2 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 1 | 2 | 0
Pneumonia (Infections and infestations) | 10 | 10 | 2 | 3
Sepsis (Infections and infestations) | 2 | 3 | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 5 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 6 | 5 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 9 | 10 | 3 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 19 | 3 | 5 | 1
Alanine aminotransferase increased (Investigations) | 13 | 6 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 13 | 9 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 6 | 10 | 0 | 0
Blood bilirubin increased (Investigations) | 19 | 11 | 3 | 2
Blood creatinine increased (Investigations) | 8 | 14 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 11 | 0 | 0
Neutrophil count decreased (Investigations) | 9 | 22 | 2 | 0
Platelet count decreased (Investigations) | 17 | 24 | 4 | 2
Weight decreased (Investigations) | 9 | 8 | 1 | 1
White blood cell count decreased (Investigations) | 6 | 14 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 20 | 21 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5 | 3 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 7 | 4 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 12 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 8 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 22 | 5 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 8 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 14 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 8 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 10 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 6 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 8 | 2 | 1
Dysgeusia (Nervous system disorders) | 5 | 6 | 0 | 0
Headache (Nervous system disorders) | 13 | 11 | 5 | 2
Presyncope (Nervous system disorders) | 3 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 5 | 5 | 1 | 3
Confusional state (Psychiatric disorders) | 5 | 5 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 6 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 4 | 2 | 1
Haematuria (Renal and urinary disorders) | 5 | 6 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 16 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 15 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 5 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 9 | 0 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 5 | 1 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3
Haematoma (Vascular disorders) | 1 | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 5 | 2 | 5
Hypotension (Vascular disorders) | 12 | 6 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT04778397/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04778397/SAP_001.pdf